CLINICAL TRIAL: NCT02726256
Title: G-CREDIT (Gangnam-Cohort for Risk Evaluation of Diabetes and Impaired Glucose Tolerance)
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2010-0195
Record Dates: First submitted 2016-03-27; First posted 2016-04-01 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes; Impaired Glucose Intolerance
Keywords: Diabetes; DM complication
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample in EDTA containing tube would be refrigerated and used in developing a new biomarker
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes and Impaired glucose Tolerance (G-CREDIT): Patients with either type 2 diabetes or impaired glucose tolerance who are older than 20 years old and have attended Gangnam Severance hospital for regular follow up.

SUMMARY:
The prevalence of type 2 diabetes has consistently increased and type 2 diabetes can cause many types of vascular complications. Diabetes develops due to glucose intolerance. Early detection and intervention in the stage of glucose intolerance makes it afford to prevent overt diabetes and its complications. This study was designed to make a cohort of korean patients with glucose intolerance to construct a long term database about clinical characteristics of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 20 years old who has visited Gangnam severance hospital since January 2007.
2. Patients with either diabetes or impaired glucose tolerance
3. Patients with at least 6 months of follow-up period

Exclusion Criteria:

1. Patients with gestational diabetes, any active stage of cancer and severe disability

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either type 2 diabetes or impaired glucose toloerance who are older than 20 years old and have attended Gangnam Severance hospital for regular follow up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-01; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Life style assessment - Past medical history - Smoking, alcohol history - Sleep, exercise, daily activity check - Diet - Reproductive status (Women only) - Socioeconomic status | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Past medical history | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Smoking, alcohol history | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Sleep, exercise, daily activity check | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Diet | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Reproductive status (Women only) | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Socioeconomic status | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Anthropometric measurements : Height, weight, waist circumference, pulse rate, blood pressure | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
SMA, TG, HDL, LDLM apoA, apoB | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
PC2hrs, HbA1C, Insulin, C-peptide (AC, PC2hr), hs-CRP | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Urine protein, albumin, creatinine | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
EKG, Neurometer, Chest PA, Abdominal sonography | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
Fundus photography, fat computed tomography | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications
HOMA-IR, HOMA-β | an expected average of 12 weeks
  Measuring above all, investigators plan to investigate how clinical parameters help to predict and prevent diabetic vascular complications

IPD SHARING:
Plan to Share IPD: Yes
This study has a plan to share data